CLINICAL TRIAL: NCT05159310
Title: A Randomized Controlled Trial Comparing Clinical Outcomes of Casting Versus Splinting in Distal Radius Fractures in Patients 60 Years and Above
Brief Title: Cast Vs Splint in Distal Radius Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/00510
Record Dates: First submitted 2021-11-09; First posted 2021-12-16 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: The study methodology will be a non-inferiority randomized controlled trial (RCT). A non-inferiority design was selected because it is unlikely that splints are superior to casts with regards to the primary outcome - final functional outcome at 12 months. Both intention-to-treat and per-protocol analyses will be performed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast (Other): Patients presenting with DRF will be screened by the attending consultant. The temporary backslab will be removed, X-rays will be obtained, and the attending consultant will discuss the treatment options. Patients who are planned for non-operative treatment and meet the inclusion criteria will be eligible for the study. The purpose and details of the study will be explained and informed consent will then be taken by the research coordinator (RC). The participants will then be randomized (using a block-randomization method) to either treatment by splint or cast. A research assistant will facilitate the randomisation process so that the RC and the treating physician remain blinded to treatment allocation.
  Interventions: Procedure: Cast vs Splint
- Splint (Other): Patients presenting with DRF will be screened by the attending consultant. The temporary backslab will be removed, X-rays will be obtained, and the attending consultant will discuss the treatment options. Patients who are planned for non-operative treatment and meet the inclusion criteria will be eligible for the study. The purpose and details of the study will be explained and informed consent will then be taken by the research coordinator (RC). The participants will then be randomized (using a block-randomization method) to either treatment by splint or cast. A research assistant will facilitate the randomisation process so that the RC and the treating physician remain blinded to treatment allocation.
  Interventions: Procedure: Cast vs Splint

INTERVENTIONS:
Procedure: Cast vs Splint — Patients presenting with DRF will be screened by the attending consultant. The temporary backslab will be removed, X-rays will be obtained, and the attending consultant will discuss the treatment options. Patients who are planned for non-operative treatment and meet the inclusion criteria will be eligible for the study. The purpose and details of the study will be explained and informed consent will then be taken by the research coordinator (RC). The participants will then be randomized (using a block-randomization method) to either treatment by splint or cast.

SUMMARY:
This study will evaluate and compare the efficacy of 2 commonly-used methods of fracture immobilisation: (1) Fiberglass cast, and (2) Thermoplastic splint. Both these devices are externally applied and provide pain relief while immobilising the fracture in an acceptable position. Casts and splints are both established devices in routine clinical use.

DETAILED DESCRIPTION:
Casts and splints are both established methods of treating DRF. Casts have been traditionally the gold standard for non-operative care of fractures, but there are distinct disadvantages such as skin rash and pruritus, malodour, skin maceration and loosening as the initial swelling subsides. Casts require specialized tools for removal and they have to be reapplied by specialized staff if the casts become loose or wet. Splints have the advantage of being removable and therefore facilitate hygiene and provide a better fit because of the adjustable straps. Splints are theoretically less rigid and patient non-compliance because of the ease of removal may result in a greater likelihood of fracture displacement. However, it is known that fractures displace even in casts and the efficacy of casts at maintaining reduction over splints has not been established. Moreover, it has been clearly shown that the elderly patients have good functional outcomes that do not correlate with the position in which the fracture heals i.e. they tolerated a large degree of fracture malunion (Arora; Egol).

The primary goal of this study is to show that there is no difference in the final functional outcome between distal radius fractures treated non-operatively with splints and casts. The secondary goals are to demonstrate: (1) splinting results in greater patient comfort and acceptance; (2) there is no significant difference in final radiographic outcomes between DRF treated with casts and splints; and (3) there is no difference in clinical outcome at the 6-month and 12-month follow-up points.

This study is clinically important for several reasons. First, patients may be encouraged to use splints instead of casts if there is no difference in functional outcome and the former provide better comfort. Second, patients may not be required to present for long (>6-month) follow-ups if it can be shown that the clinical improvement plateaus at 6 months after injury. This is consistent with our aim to improve patients' overall quality of life after musculoskeletal injuries and forms a core component of functional ageing.

ELIGIBILITY:
Inclusion Criteria:

* Closed DRF in patients > 60 years
* Presenting to HRMC within 10 days of injury
* Isolated injury
* With or without M&R performed in EMD
* Declined surgical fixation after appropriate discussion

Exclusion Criteria:

* Wounds - skin tears, bad abrasions, open fracture
* Ulnar fracture > styloid
* Other MSK / non-MSK injuries
* Bilateral fractures
* Prior wrist fractures / wrist surgery
* Other upper limb conditions affecting function (e.g. CVA)
* Cognitive impairment
* Allergy to plaster or fiberglass

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Splinting results in Quick Disabilities of Arm, Shoulder, Hand (QuickDASH) scores that are not poorer as compared to casting | 12 months
  The resultant score is reported on a scale of 0 to 100, where 0 represents no disability and 100 represents total disability.
  Splinting in patients ≥60 years with distal radius fracture (DRF) results in 12-month QuickDASH scores that are significantly inferior compared to scores in patients treated in cast.
  The alternate hypothesis is that splinting results in 12-month QuickDASH scores that are not significantly inferior compared to casting in this group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Soumen Das De, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Records for all participants, including all source documentation (containing evidence to study eligibility, history and physical findings, results of consultations etc) as well as IRB records and other regulatory documentation will be retained by the principal investigator via the following means:
  * Electronic records will be kept on an encrypted hard drive
  * Hardcopy data will be stored in a locked cabinets in the office of the principal investigator and accessed only by the principal investigator, co-investigators or study administrators.